CLINICAL TRIAL: NCT03198611
Title: Early Reversibility of Diastolic Disfunction as a Prognostic Factor in Septic Shock
Brief Title: Reversibility of Diastolic Disfunction in Septic Shock
Acronym: REPRISS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Other Study IDs: IIBSP-REP-2017-30
Record Dates: First submitted 2017-06-16; First posted 2017-06-26 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Diastolic Dysfunction; Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal function: No systolic dysfunction No diastolic dysfunction No right ventricular dysfunction
  Interventions: Diagnostic Test: Echocardiography
- Left ventricular systolic dysfunction: Left ventricular ejection fraction < 50%
  Interventions: Diagnostic Test: Echocardiography
- Left ventricular diastolic dysfunction: Classification according to:
  * Mitral lateral annulus e' in tissue Doppler < 10 cm/s
  * American society of echocardiography (ASE) criteria 2009
  * ASE criteria 2016
  Interventions: Diagnostic Test: Echocardiography
- Right ventricular dysfunction: Tricuspid annulus plane systolic excursion < 17 cm
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Usual echocardiographic studies in patients suffering septic shock

SUMMARY:
Objectives: To study the prognostic value of the evolution of diastolic function according to fluid balance in patients admitted to the ICU with a diagnosis of septic shock, in terms of mortality (ICU and hospital) and mortality at 90 days.

2.4. Secondary objectives: A) Incidence and reversibility of myocardial dysfunction (left ventricular systolic and diastolic) in septic shock.

B) Incidence and reversibility of diastolic dysfunction according to the echocardiographic criterion used.

C) Incidence and reversibility of right ventricular systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU with diagnosis of septic shock, and stay longer than 48h

Exclusion Criteria:

* No echocardiographic window
* Fatal prognosis with do not resuscitate orders at admission
* Previous history of Ischemic cardiomyopathy
* Valvular prosthesis
* Advanced degree of valvular disorder
* Advanced degree of pericardial effusion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with diagnosis of septic shock, and stay longer than 48h
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Mortality at 90 days | 90 days
  Dead at 90 days

SECONDARY OUTCOMES:
ICU mortality | 90 days
  Dead in ICU
In hospital mortality | 90 days
  Dead in hospital
Incidence of myocardial disfunction | During the first 24 hours of ICU admission
  According to the criteria specified at groups section
Change in incidence of diastolic dysfunction | From first 24 hours of ICU admission until 48h, 72h and 7 days from admission
  Change in incidence of diastolic dysfunction according to the different criteria used.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital del Vall d´Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Suarez JC, Lopez P, Mancebo J, Zapata L. Diastolic dysfunction in the critically ill patient. Response from the authors. Med Intensiva. 2017 Apr;41(3):198. doi: 10.1016/j.medin.2016.12.008. Epub 2017 Mar 3. No abstract available. English, Spanish. PMID 28262372
- [Background] Mahjoub Y, Benoit-Fallet H, Airapetian N, Lorne E, Levrard M, Seydi AA, Amennouche N, Slama M, Dupont H. Improvement of left ventricular relaxation as assessed by tissue Doppler imaging in fluid-responsive critically ill septic patients. Intensive Care Med. 2012 Sep;38(9):1461-70. doi: 10.1007/s00134-012-2618-9. Epub 2012 Jun 21. PMID 22717694
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Alexandru Popescu B, Waggoner AD; Houston, Texas; Oslo, Norway; Phoenix, Arizona; Nashville, Tennessee; Hamilton, Ontario, Canada; Uppsala, Sweden; Ghent and Liege, Belgium; Cleveland, Ohio; Novara, Italy; Rochester, Minnesota; Bucharest, Romania; and St. Louis, Missouri. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2016 Dec;17(12):1321-1360. doi: 10.1093/ehjci/jew082. Epub 2016 Jul 15. No abstract available. PMID 27422899